## **INFORMED CONSENT**

Name of the Study:

"Usefulness of Oscillometry in Assessing the Effectiveness of Inhaled Corticosteroides in Patients With COPD Exacerbator Phenotype"

This form must be provided by one of the study's pulmonologists before the

| analysis is performed. | |
|---------------------------------------------------------|---|
| <u> </u> | |
| <patient's full="" name=""></patient's> | |
| I have read the information sheet that was given to me. | |
| I have been able to ask questions about the study. | |
| I have received sufficient information about the study. | |
| I have spoken with: | |
| Study researcher | _ |
| I understand that my participation is voluntary. | |
| I understand that I may withdraw from the study: | |
| 1st Whenever you want. | |
| 2nd Without having to give explanations. | |
| 3rd Without this affecting my medical care. | |

Distribution: original to the researcher, copy to the patient.